CLINICAL TRIAL: NCT04110691
Title: Impact of Stent Length and Diameter on Short Term Outcomes in Patients With ST Segment Elevation Myocardial Infarction Undergoing Primary PCI.
Brief Title: Impact of Stent Length and Diameter on Patients Undergoing Primary PCI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Deyaa, Principal investigator, Assiut University
Other Study IDs: coronary stents
Record Dates: First submitted 2019-09-28; First posted 2019-10-01 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the study is to evaluate the Impact of coronary stent length and/or diameter in patients with ST segment myocardial infarction undergoing primary PCI, on Short term clinical outcomes.

DETAILED DESCRIPTION:
* ST segment elevation myocardial infarction is serious condition to the blood supply to the heart muscle. Rapid reperfusion of the ischemic myocardium using percutaneous coronary intervention (PCI) is the standard treatment for acute myocardial infarction (MI) to rescue the ischemic myocardium and reduce infarction size.
* There are two types of stents:

  1. Drug-eluting stent which achieving local drug delivery to the injured blood vessel at the time of intervention, a drug is released from a polymer coating or loaded directly onto the stent (2). This is the best one.
  2. Bare metal stent is the old one and not effective as DES in reducing vascular restenosis by suppressing smooth muscle cell (SMC) proliferation.
* The management of long coronary lesions by percutaneous coronary intervention (PCI) has become increasingly important because of the rising incidence of long or complex lesions in aging populations (3) Stent length has been considered as an important predictor of adverse events after PCI. The exact impact of lesion length on the short- and long-term clinical outcomes of DES implantations is not clear yet.
* Myocardial necrosis complicates one-third of percutaneous coronary intervention (PCI) and may adversely affect the outcome(4)

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST segment myocardial infarction who are eligible for PCI.
* All categories (all age groups and both sex groups)

Exclusion Criteria:

* Patients with previous PCI.
* Patients of ectatic lesions.
* Patients with with multi vessel disease and suitable for CABG.
* Patients with complex lesions including bifurcational lesions and LM stenting.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ST segment elevation myocardial infarction undergoing primary PCI
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-01-28 (Estimated)

PRIMARY OUTCOMES:
prognosis of patients with ST segment myocardial infarction undergoing primary PCI | 3 months
  prognosis will be measured with ECG and ECHO

CONTACTS AND LOCATIONS:
Overall Officials: Nada Deyaa, Principal Investigator — Assiut University